CLINICAL TRIAL: NCT03108690
Title: Therapeutic Drug Monitoring and Continuous Infusion of Beta-lactam Antibiotics in Patients With Bacteraemia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Logistics
Sponsor: Sara Thønnings (Other)
Responsible Party: Sponsor-Investigator, Sara Thønnings, MD, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-768
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Bacteremia
Keywords: Therapeutic drug monitoring; Continuous infusion; Beta-lactam; Antibiotics; Bacteraemia
MeSH Terms: conditions — Bacteremia; Toxemia | interventions — Penicillin G; Ampicillin; Dicloxacillin; Piperacillin, Tazobactam Drug Combination; Cefuroxime; Meropenem

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TDM and CI. (Experimental): Continuous infusion of beta-lactam antibiotics. Therapeutic drug monitoring of beta-lactam antibiotics.
  Interventions: Drug: Continuous infusion of beta-lactam antibiotics .; Other: Therapeutic drug monitoring of beta-lactam antibiotics.
- Control (No Intervention): Beta-lactam antibiotics given as intermittent infusion. Samples of serum concentration of beta-lactam will be collected for comparison, but blinded during the study.

INTERVENTIONS:
Drug: Continuous infusion of beta-lactam antibiotics . — Beta-lactam antibiotic will be administered as continous infusion.
  Other Names: Benzylpenicillin; Ampicillin; Dicloxacillin; Piperacillin/tazobactam; Cefuroxime; Meropenem
  Arms: TDM and CI.
Other: Therapeutic drug monitoring of beta-lactam antibiotics. — Dosage of beta-lactam antibiotics will be adjusted according to serum concentration.
  Arms: TDM and CI.

SUMMARY:
The study investigates whether Therapeutic Drug Monitoring (TDM) and continuous infusion (CI) of beta-lactam antibiotics optimises target concentrations in patients with bacteraemia.

ELIGIBILITY:
Inclusion Criteria:

* Have a positive blood culture.
* Undergo treatment with either intravenous penicillin, ampicillin, piperacillin/tazobactam, dicloxacillin, cefuroxime or meropenem.
* Hospitalised at Hvidovre University Hospital.
* Age ≥ 18.
* Able to understand and give informed consent.
* Included in the study within 24 hours after the final positive blood culture answer.

Exclusion Criteria:

* Positive blood culture is interpreted as contamination.
* The patient dies before the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Target concentrations. | 30 days after intervention.
  Serum concentrations within the target values for intervention. Following beta-lactams is included in the study: Benzylpenicillin, ampicillin, dicloxacillin, piperacillin/tazobactam, cefuroxime and meropenem.

SECONDARY OUTCOMES:
Morbidity. | 30 days after intervention.
  Diagnoses compared between the two arms.
Number of days until medically discharged. | 30 days after intervention.
  Number of days until medically discharged compared between the two arms.
Failed antibiotic treatments. | 30 days after intervention.
  Adding an additional antibiotic and/or change to a different antibiotic (not including a more narrow spectrum antibiotic) compared between the two arms.
Amount of antibiotic used. | 30 days after intervention.
  Defined daly doses of antibiotic therapy compared between the two arms.
Antibiotic side effects and complications. | 30 days after intervention.
  The severity of bacteraemia, mechanical ventilation and start-up of dialysis compared between the two arms. Growth of antibiotic-associated pathogenic in patient material compared between the two arms.
Mortality. | 30 days after intervention.
  30-day mortality compared between the two arms.
Number of participants with abnormal clinical data and/or abnormal laboratory values. | 30 days after intervention.
  Clinical data includes height, weight, heart rate, blood pressure, respiratory rate, Glasgow Coma Scale score, body temperature, fous of infection, the severity of bacteraemia, dialysis and laboratory values includes hemoglobin, white blood cells, neutrophils, thrombocytes, C-reactive protein, sodium, potassium, creatinine, albumin, lactate dehydrogenase, alanine amino transferase and lactate. Both will be compared between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Thønnings, MD, Principal Investigator — Hvidovre University Hospital